CLINICAL TRIAL: NCT01516567
Title: Intergroup Trial for Children or Adolescents With B-Cell NHL or B-AL: Evaluation of Rituximab Efficacy and Safety in High Risk Patients - Phase II Trial of DA-EPOCH-Rituximab in PMLBL
Brief Title: Intergroup Trial for Children or Adolescents With Primary Mediastinal Large B-Cell Lymphoma: DA-EPOCH-Rituximab Evaluation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inter B-NHL Ritux 2010 Phase 2; 2010-019224-31 (EudraCT Number); NCT01595048 (obsolete NCT alias)
Record Dates: First submitted 2012-01-19; First posted 2012-01-25 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Primary Mediastinal Large B Cell Lymphoma
MeSH Terms: interventions — Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DA-EPOCH-R (Experimental): 6 courses of Dose Adjusted-EPOCH-Rituximab
  Interventions: Drug: Etoposide, Doxorubicin, Vincristine, Cyclophosphamide, Rituximab

INTERVENTIONS:
Drug: Etoposide, Doxorubicin, Vincristine, Cyclophosphamide, Rituximab — 6 courses of Dose Adjusted-EPOCH-Rituximab Rituximab 375 mg/m² i.v.: one injection at each of the 6 courses of EPOCH.

SUMMARY:
Phase II trial to determine the efficacy of Dose Adjusted-EPOCH-Rituximab regimen in children and adolescent with primary mediastinal large B cell lymphoma in terms of event free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Primary Mediastinal Large B-Cell Lymphoma (PMLBL).
* PMLBL without central nervous system (CNS) involvement.
* 6 months to less than 18 years of age at the time of consent.
* Males and females of reproductive potential must agree to use an effective contraceptive method during the treatment, and after the end of treatment: during twelve months for women, taking into account the characteristics of rituximab
* Complete initial work-up within 8 days prior to treatment that allows definite staging.
* Able to comply with scheduled follow-up and with management of toxicity.
* Signed informed consent from patients and/or their parents or legal guardians

Exclusion Criteria:

* Follicular lymphoma, mucosa-associated lymphoid tissue (MALT) and nodular marginal zone
* PMLBL patients with CNS involvement
* Patients with congenital immunodeficiency, chromosomal breakage syndrome, prior organ transplantation, previous malignancy of any type, or known positive HIV serology.
* Evidence of pregnancy or lactation period.
* There will be no exclusion criteria based on organ function.
* Past or current anti-cancer treatment except corticosteroids during less than one week.
* Tumor cell negative for CD20
* Prior exposure to rituximab.
* Severe active viral infection, especially hepatitis B.
* Hepatitis B carrier status history of hepatitis B virus (HBV) or positive serology.
* Participation in another investigational drug clinical trial.
* Patients who, for any reason, are not able to comply with the national legislation.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Event free survival | 36 months
  Minimum time to death from any cause, presence of viable cells in residue after 6th DA-EPOCH course, relapse, progressive disease, or second malignancy measured from registration.

SECONDARY OUTCOMES:
Survival | 5 years
  Overall survival
Acute toxicity | 6 months
  Acute toxicity during treatment according to NCI-CTC V4
Long term toxicity | 5 years
  Long term toxicity, especially immune reconstitution, cardiac toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PATTE, MD, Study Chair — Institut Gustave Roussy, Villejuif, FRANCE; Thomas GROSS, MD, Study Chair — Children's Oncology Group, USA
Locations (9):
- University Hospitals Leuven, Leuven, Belgium
- Children Oncology Group Operations centres, Monrovia, Canada
- Gustave Roussy, Villejuif, France
- 2nd Dept. of Pediatrics Semmelweis Univ., Budapest, Hungary
- Associazione Italiana di Ematologia ed Oncologia Pediatrica, Padua, Italy
- Emma Children's Hospital, Amsterdam, Netherlands
- Rectorat of Medical University, Wroclaw, Poland
- Sociedad Española de Hematología y Oncología Pediátricas, Valencia, Spain
- University of Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Burke GAA, Minard-Colin V, Auperin A, Alexander S, Pillon M, Delgado R, Zsiros J, Uyttebroeck A, Dartigues P, Miles RR, Kazanowska B, Chiang AK, Haouy S, Bollard CM, Csoka M, Wheatley K, Barkauskas DA, Adamson PC, Vassal G, Patte C, Gross TG. Dose-Adjusted Etoposide, Doxorubicin, and Cyclophosphamide With Vincristine and Prednisone Plus Rituximab Therapy in Children and Adolescents With Primary Mediastinal B-Cell Lymphoma: A Multicenter Phase II Trial. J Clin Oncol. 2021 Nov 20;39(33):3716-3724. doi: 10.1200/JCO.21.00920. Epub 2021 Sep 27. PMID 34570655
- See also: Institute Gustave Roussy web site — http://www.igr.fr